CLINICAL TRIAL: NCT00641251
Title: Global Randomized Prospective Study of Intensive Medical Management of Type 2 Diabetes, With and Without Gastric Bypass Surgery
Brief Title: DSS: Diabetes Surgery Study - Intensive Medical Management of Type 2 Diabetes, With and Without Gastric Bypass Surgery
Acronym: DSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AS07008
Record Dates: First submitted 2008-02-13; First posted 2008-03-24 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Type 2 Diabetes; Cardiovascular Disease
Keywords: T2 Diabetes; Type 2 diabetes CVD event rates and mortality
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): intensive medical management
  Interventions: Other: intensive medical management
- 2 (Active Comparator): Roux-en-Y gastric bypass with intensive medical management
  Interventions: Other: RYGB & IMM

INTERVENTIONS:
Other: intensive medical management — IMM will include rigorous lifestyle modification for weight loss and stepped pharmacologic treatment consistent with standard of care for diabetes and other CVD risk factors.
  Arms: 1
Other: RYGB & IMM — Roux-en-Y gastric bypass Surgery combined with intensive medical management
  Arms: 2

SUMMARY:
The present study is the first stage of a research program whose ultimate goal is to conduct a randomized clinical trial involving type 2 diabetics with BMI from 30.0 to 39.9 kg/m2. This program will determine the relative effectiveness of RYGB combined with intensive medical management (IMM), versus IMM alone, in reducing CVD event rates and mortality in patients with poorly controlled diabetes. IMM will include rigorous lifestyle modification for weight loss and stepped pharmacologic treatment for diabetes and other CVD risk factors. The proposed study is a randomized trial which will provide an assessment of the efficacy of treatment, in reducing CVD risk factors and also assessing the feasibility, cost, and safety of a larger trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30 to 67 years at eligibility visit.
2. Diagnosed with T2DM at least 6 months prior to enrollment, under the active care of a doctor for at least the six months prior to enrollment, and HbA1c ≥ 8.0 %.
3. Body Mass Index (BMI) ≥ 30.0 kg/m2 and ≤ 39.9 kg/m2 at eligibility visit.
4. Willingness to accept random assignment to either treatment group.
5. Expect to live or work within approximately one hour's traveling time from the study clinic for the duration of the two-year trial.
6. Willingness to comply with the follow-up protocol and successful completion of the run-in (described below).
7. Written informed consent.

Exclusion Criteria:

1. Cardiovascular event (myocardial infarction, acute coronary syndrome, coronary artery angioplasty or bypass, stroke) in the past six months.
2. Current evidence of congestive heart failure, angina pectoris, or symptomatic peripheral vascular disease.
3. Cardiac stress test indicating that surgery or IMM would not be safe.
4. Pulmonary embolus or thrombophlebitis in the past six months.
5. Cancer of any kind (except basal cell skin cancer or cancer in situ) unless documented to be disease-free for five years.
6. Significant anemia (hemoglobin 1.0 g or more below normal range) or history of coagulopathy.
7. Serum creatinine ≥ 1.5 mg/dl.
8. HbA1c > 14.0%.

Ages: 30 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
HbA1c < 7.0% | 12 Months
Systolic blood pressure < 130 mm Hg | 12 Months
LDL cholesterol < 100 mg/dl | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Sayeed Ikramuddin, MD, Principal Investigator — University of Minnesota
Locations (5):
- United States (3):
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University, New York, New York
- Taiwan (2):
  - Min-Sheng General Hospital, Taipei
  - National Taiwan University Hospital, Taipei

REFERENCES:
- [Derived] Ikramuddin S, Korner J, Lee WJ, Thomas AJ, Connett JE, Bantle JP, Leslie DB, Wang Q, Inabnet WB 3rd, Jeffery RW, Chong K, Chuang LM, Jensen MD, Vella A, Ahmed L, Belani K, Billington CJ. Lifestyle Intervention and Medical Management With vs Without Roux-en-Y Gastric Bypass and Control of Hemoglobin A1c, LDL Cholesterol, and Systolic Blood Pressure at 5 Years in the Diabetes Surgery Study. JAMA. 2018 Jan 16;319(3):266-278. doi: 10.1001/jama.2017.20813. PMID 29340678
- [Derived] Chong K, Ikramuddin S, Lee WJ, Billington CJ, Bantle JP, Wang Q, Thomas AJ, Connett JE, Leslie DB, Inabnet WB 3rd, Jeffery RW, Sarr MG, Jensen MD, Vella A, Ahmed L, Belani K, Schone JL, Olofson AE, Bainbridge HA, Laqua PS, Korner J, Chuang LM. National Differences in Remission of Type 2 Diabetes Mellitus After Roux-en-Y Gastric Bypass Surgery-Subgroup Analysis of 2-Year Results of the Diabetes Surgery Study Comparing Taiwanese with Americans with Mild Obesity (BMI 30-35 kg/m2). Obes Surg. 2017 May;27(5):1189-1195. doi: 10.1007/s11695-016-2433-4. PMID 27783367
- [Derived] Ikramuddin S, Korner J, Lee WJ, Bantle JP, Thomas AJ, Connett JE, Leslie DB, Inabnet WB 3rd, Wang Q, Jeffery RW, Chong K, Chuang LM, Jensen MD, Vella A, Ahmed L, Belani K, Olofson AE, Bainbridge HA, Billington CJ. Durability of Addition of Roux-en-Y Gastric Bypass to Lifestyle Intervention and Medical Management in Achieving Primary Treatment Goals for Uncontrolled Type 2 Diabetes in Mild to Moderate Obesity: A Randomized Control Trial. Diabetes Care. 2016 Sep;39(9):1510-8. doi: 10.2337/dc15-2481. Epub 2016 Jun 16. PMID 27311493
- [Derived] Ikramuddin S, Billington CJ, Lee WJ, Bantle JP, Thomas AJ, Connett JE, Leslie DB, Inabnet WB 3rd, Jeffery RW, Chong K, Chuang LM, Sarr MG, Jensen MD, Vella A, Ahmed L, Belani K, Schone JL, Olofson AE, Bainbridge HA, Laqua PS, Wang Q, Korner J. Roux-en-Y gastric bypass for diabetes (the Diabetes Surgery Study): 2-year outcomes of a 5-year, randomised, controlled trial. Lancet Diabetes Endocrinol. 2015 Jun;3(6):413-422. doi: 10.1016/S2213-8587(15)00089-3. Epub 2015 May 12. PMID 25979364
- [Derived] Ikramuddin S, Korner J, Lee WJ, Connett JE, Inabnet WB, Billington CJ, Thomas AJ, Leslie DB, Chong K, Jeffery RW, Ahmed L, Vella A, Chuang LM, Bessler M, Sarr MG, Swain JM, Laqua P, Jensen MD, Bantle JP. Roux-en-Y gastric bypass vs intensive medical management for the control of type 2 diabetes, hypertension, and hyperlipidemia: the Diabetes Surgery Study randomized clinical trial. JAMA. 2013 Jun 5;309(21):2240-9. doi: 10.1001/jama.2013.5835. PMID 23736733